CLINICAL TRIAL: NCT01551264
Title: Duration of Brace Wear in Clubfoot Treatment - A Prospective Randomized Trail
Brief Title: Duration of Brace Wear in Clubfoot Treatment - A Prospective Randomized Trial
Acronym: FAB24
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201110158
Record Dates: First submitted 2012-03-07; First posted 2012-03-12 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Isolated Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4-Year Bracing Arm (Other): This group has been randomized to 4 years of bracing after correction of clubfoot using the Ponseti Method.
  Interventions: Device: Foot Abduction Brace (FAB)
- 2-Year Bracing Arm (Other): This group has been randomized to 2 years of bracing after correction of clubfoot using the Ponseti Method.
  Interventions: Device: Foot Abduction Brace (FAB)

INTERVENTIONS:
Device: Foot Abduction Brace (FAB) — After clubfoot correction, the participants will wear the FAB 23 hours/day for 3 months and then wean to naps and nighttime (8-12 hours/day) for either 2 or 4 years depending on which arm they are in.

SUMMARY:
The goal of this multi-center, randomized, controlled trial is to evaluate the effectiveness of a 2 year versus 4 year bracing protocol in preventing isolated clubfoot recurrence within the first year post-treatment, and to evaluate factors associated with recurrence in isolated clubfoot.

DETAILED DESCRIPTION:
The study is based on the hypothesis that prolonged bracing will reduce clubfoot recurrence. In addition to bracing length, the study will determine if other factors in addition to duration of brace wear are associated with recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Subject < 1 year of age when treatment initiated at local site
* Confirmed diagnosis of Isolated Clubfoot
* At least one foot demonstrates fixation of the foot in equinus, forefoot adduction, cavus and hindfoot varus
* Deformity was present at birth

Exclusion Criteria:

* Previous foot abduction bracing
* Previous surgical correction (excluding Tenotomy)
* Dysmorphic features, additional anomalies (i.e. congenital heart disease, hypospadias, a genetic syndrome), or developmental delay
* Neurologic cause for clubfoot (i.e. myelomeningocele or sacral agenesis)

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Dobbs, MD, Principal Investigator — Washington University School of Medicine
Locations (7):
- United States (7):
  - Shriners Hospital for Children, Sacramento, California
  - Nemours Children's Hospital, Orlando, Florida
  - Shriners Hospital for Children, Lexington, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - Shriners Hospital for Children, St Louis, Missouri
  - Shriners Hospital for Children, Portland, Oregon
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Result] Dobbs MB, Frick SL, Mosca VS, Raney E, VanBosse HJ, Lerman JA, Talwalkar VR, Steger-May K, Gurnett CA. Design and descriptive data of the randomized Clubfoot Foot Abduction Brace Length of Treatment Study (FAB24). J Pediatr Orthop B. 2017 Mar;26(2):101-107. doi: 10.1097/BPB.0000000000000387. PMID 27632641

RESULTS

PARTICIPANT FLOW:
Groups:
- 4-Year Bracing Arm: This group has been randomized to 4 years of bracing after correction of clubfoot using the Ponseti Method.
  Foot Abduction Brace (FAB): After clubfoot correction, the participants will wear the FAB 23 hours/day for 3 months and then wean to naps and nighttime (8-12 hours/day) for 4 years.
- 2-Year Bracing Arm: This group has been randomized to 2 years of bracing after correction of clubfoot using the Ponseti Method.
  Foot Abduction Brace (FAB): After clubfoot correction, the participants will wear the FAB 23 hours/day for 3 months and then wean to naps and nighttime (8-12 hours/day) for 2 years.
Period: Overall Study
Arm/Group | 4-Year Bracing Arm | 2-Year Bracing Arm
Started (Enrolled and Randomized) | 70 | 69
Started Bracing | 69 | 67
Data for at Least One Follow-up After Brace Discontinuation Ascertained | 44 (Attended at least one visit within one year after discontinuing bracing) | 55 (Attended at least one visit within one year after discontinuing bracing)
Completed (One year follow-up after brace discontinuation ascertained) | 38 (Attended 60 month follow-up visit) | 41 (Attended 36 month follow-up visit)
Not Completed | 32 | 28

BASELINE CHARACTERISTICS:
Population: Baseline participants represent the number of participants enrolled and randomized. However, participant could drop out of the study prior to starting the bracing treatment due to eligibility changes or site discontinuation.
Groups:
- Total: Total of all reporting groups
Arm/Group | 4-Year Bracing Arm | 2-Year Bracing Arm | Total
Number analyzed (Participants) | 70 | 69 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 70 | 69 | 139
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] — Age at study consent
  Months | 1.8 (1.7) | 1.8 (1.5) | 1.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 41
  Male | 52 | 46 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 4 | 8
  White | 57 | 59 | 116
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 70 | 69 | 139
Measure Description: Laterality of isolated clubfoot at enrollment [Count of Participants; unit: Participants]
  Unilateral | 35 | 35 | 70
  Bilateral | 35 | 34 | 69
Family history of clubfoot in first-degree relative [Count of Participants; unit: Participants]
  Presence | 9 | 10 | 19
  Absence | 61 | 59 | 120

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Recurrence-Free Survival Probability for Clubfoot Affected Limbs
Description: Kaplan-Meier recurrence-free survival probability for each limb affected by clubfoot up to 1 year after bracing is discontinued. For patients with bilateral clubfoot, each limb was assessed. Bilateral patients contribute data for both limbs and unilateral patients contribute data for the affected limb. Recurrence is defined as the development of any of the following deformities in isolation or in combination that require repeat cast application or surgical intervention: hindfoot varus, ankle equinus, midfoot adduction, midfoot cavus, or forefoot pronation. Clubfoot recurrence was determined by the local Principal Investigator.
Time Frame: From end of bracing treatment until the earliest recurrence up to 1 year (allowing for per-protocol visit window of 1.2 years) after the assigned treatment (2- or 4-year bracing) is discontinued.
Population: For patients with bilateral clubfoot, each limb was assessed. Bilateral patients contribute data for both limbs and unilateral patients contribute data for the affected limb. Analysis includes limbs from participants who started bracing and attended at least one visit within one year after discontinuing bracing.
Measure: Number (95% Confidence Interval); unit: survival probability
Units Other Than Participants: limb
Arm/Group | 4-Year Bracing Arm | 2-Year Bracing Arm
Number analyzed (Participants) | 44 | 55
Number analyzed (limb) | 65 | 82
survival probability | 0.81 [0.70 to 0.95] | 0.65 [0.52 to 0.80]
Statistical Analysis 1: Comparison: 4-Year Bracing Arm vs 2-Year Bracing Arm; Test type: Other — P-value by chi-square comparing the Kaplan-Meier recurrence-free survival probability at 1.2 years post treatment with robust estimate of standard error due to the a priori assumption that data from bilateral limbs are correlated; p = 0.03, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events for each participant were evaluated from participant randomization to the last study visit attended. For participants that completed the study, the last study visit is 60 months after brace fitting. For participants that did not complete the study, the last study visit is the final study visit that the participant attended.
Description: An adverse event is any new untoward medical occurrence or worsening of a preexisting medical condition that occurs in association with study procedures (consent process, questionnaires, loss of protected health information) or treatment reaction in excess of expectation. Serious adverse events require extensive or urgent intervention/corrective action, pose immediate threat of harm, or death. Relatedness is defined as: clearly related, likely related, possibly related, or clearly not related.
Arm/Group | 4-Year Bracing Arm | 2-Year Bracing Arm
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/69
Other Adverse Events (participants affected / at risk) | 0/70 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT01551264/Prot_SAP_000.pdf